CLINICAL TRIAL: NCT07341100
Title: A Multicenter, Open-label Clinical Study to Evaluate the Preliminary Efficacy of SKB264 and the Effect of Clarithromycin, a Potent CYP3A Inhibitor, on the Pharmacokinetics of SKB264 in Patients With Ovarian Epithelial Cancer
Brief Title: Study to Evaluate the Preliminary Efficacy of SKB264 and the Effect of Clarithromycin on the PK of SKB264 in OC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-Ⅱ-19
Record Dates: First submitted 2025-12-18; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Clarithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SKB264+clarithromycin (Experimental): Cycle 1 will be for drug-drug interaction (DDI) assessment participants received SKB264 and clarithromycin .Thereafter, participants will receive SKB264 monotherapy
  Interventions: Drug: SKB264; Drug: Clarithromycin

INTERVENTIONS:
Drug: SKB264 — 4 mg/kg, administered once every 2 weeks (Q2W) by intravenous infusion. It will be administered on Day 1 and Day 17 of Cycle 1, and from Cycle 2 onwards, on Day 1 and Day 15 of each 4-week cycle.
Drug: Clarithromycin — 500 mg administered orally, twice daily (BID) from Day 14 to Day 29 of Cycle 1.

SUMMARY:
This is a multicenter, open-label study to evaluate the preliminary efficacy of SKB264 and the effect of clarithromycin on the PK of SKB264 in patients with ovarian epithelial cancer.

DETAILED DESCRIPTION:
Cycle 1 will be for drug-drug interaction (DDI) assessment. Thereafter, participants will receive SKB264 monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Females, ≥ 18 and ≤ 75 years of age at the time of signing the informed consent form (ICF).
2. Patients with histologically or cytologically confirmed recurrent ovarian epithelial cancer (including fallopian tube cancer or primary peritoneal cancer).
3. Able to provide tumor tissue samples.
4. At least one measurable lesion.
5. ECOG performance status score of 0 or 1.
6. Life expectancy ≥ 12 weeks.
7. Adequate bone marrow, liver, kidney, and coagulation function.
8. Female participants of childbearing potential must agree to use effective medical contraception from the time of signing the ICF until 6 months after the last dose.
9. The participant voluntarily agrees to participate in the study, signs the ICF, and is able to comply with the protocol-specified visits and relevant procedures.

Exclusion Criteria:

1. Participants with local recurrence who are suitable for surgery.
2. Participants who have previously undergone bone marrow radiation.
3. Ovarian cancer, fallopian tube cancer, or primary peritoneal cancer of non-epithelial origin, or other pathological types.
4. Participants with known brain metastases.
5. History of other malignancies within 3 years before the first administration.
6. There are serious cardiovascular and cerebrovascular diseases or cardiovascular and cerebrovascular risk factors.
7. Uncontrolled systemic disease as judged by the investigator.
8. History of (non-infectious) interstitial lung disease (ILD) or non-infectious pneumonitis requiring steroid therapy.
9. Documented severe dry eye syndrome, severe meibomian gland disease and/or blepharitis, or a history of severe corneal disorder that prevents/delays corneal healing.
10. Patients with serious pulmonary function impairment due to lung disease.
11. Participants with active chronic inflammatory bowel disease, gastrointestinal obstruction, severe ulcer, gastrointestinal perforation, abdominal abscess, or acute gastrointestinal hemorrhage.
12. Active gastrointestinal disease or other conditions significantly affecting the absorption, distribution, metabolism, or excretion of the oral study drug .
13. Risk of developing an esophagotracheal fistula or esophagopleural fistula, or tumor invasion or compression of surrounding vital organs and blood vessels with associated symptoms.
14. Toxicities from prior anti-tumor therapy not recovering to ≤ Grade 1.
15. Subjects with known active pulmonary tuberculosis.
16. Known history of allogeneic organ transplant and allogeneic hematopoietic stem cell transplant.
17. Active hepatitis B or hepatitis C.
18. Positive human immunodeficiency virus (HIV) test or a history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection.
19. Known hypersensitivity to any study drug or any of its components , or known severe hypersensitivity reactions to other biological agents.
20. Major surgery within 4 weeks before the first dose or expected to require major surgery during the study.
21. Serious infection within 4 weeks before the first dose.
22. Prior treatment with TROP2-targeted drug therapy or prior treatment with another topoisomerase I inhibitor as the toxin.
23. Have received any drugs that can affect CYP3A enzyme activity within 2 weeks before the first dose or within 5 half-lives of the known drug.
24. Have received any systemic anti-tumor therapy such as chemotherapy, radiotherapy , immunotherapy, targeted therapy, or biological therapy within 4 weeks before the first dose or within 5 half-lives of the known drug.
25. Have received treatment with approved traditional Chinese medicine preparations with anti-tumor indications within 2 weeks before the first dose.
26. Have received a live vaccine within 4 weeks before the first dose, or plan to receive a live vaccine during the study.
27. Any disease requiring systemic glucocorticoid therapyor other immunosuppressive drugs within 2 weeks before the first dose.
28. Participants who are currently participating in other clinical studies and receiving study drug.
29. Pregnant or lactating women.
30. Participants whose condition deteriorates rapidly before the first dose.
31. Presence of local or systemic diseases caused by non-malignant tumors.
32. Any condition that, in the opinion of the investigator, may interfere with the evaluation of the study drug or the participant's safety or the interpretation of the study results, or any other condition that the investigator deems inappropriate for participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy Endpoint | From the date of first administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Objective response rate (ORR) assessed by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Maximum observed plasma concentration (Cmax)of SKB264-ADC,SKB264-TAB and free KL610023 | The first cycle lasts for 30 days each day, and the first day of the second, third, sixth, and twelfth cycles（Starting from the second cycle, each cycle is 28 days ），up to approximately 12 months
  To assess the pharmacokinetic (PK) profile of SKB264
Area under plasma/serum concentration-time curve from zero to 13 day（AUC0-13d）of SKB264-ADC,SKB264-TAB and free KL610023 | The first cycle lasts for 30 days each day, and the first day of the second, third, sixth, and twelfth cycles（Starting from the second cycle, each cycle is 28 days ），up to approximately 12 months
  To assess the pharmacokinetic (PK) profile of SKB264
Area under plasma/serum concentration-time curve from zero to infinity（AUC0-∞）of SKB264-ADC, SKB264-TAB, and free KL610023 | The first cycle lasts for 30 days each day, and the first day of the second, third, sixth, and twelfth cycles（Starting from the second cycle, each cycle is 28 days ），up to approximately 12 months
  To assess the pharmacokinetic (PK) profile of SKB264